CLINICAL TRIAL: NCT05213039
Title: Validity and Reliability of the Timed 360° Turn Test in Children With Cerebral Palsy
Brief Title: Validity and Reliability of the the Timed 360° Turn Test
Acronym: cp
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Assistant Proffessor, Kahramanmaras Sutcu Imam University
Other Study IDs: KSUFTR1
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy; Gait, Spastic; Gait Disorders in Children; Diplegic Cerebral Palsy; Hemiplegic Cerebral Palsy
Keywords: Cerebral Palsy; the timed 360° turn test; validity; reliability
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Children with diparetic and hemiparetic cerebral palsy: 1/Children with diparetic and hemiparetic cerebral palsy whose Gross Motor Function Classification System (GMFCS) Level ≤ 2 will be evaulated by two different observers.
  Interventions: Other: assessments

INTERVENTIONS:
Other: assessments — All of the children with cerebral palsy will be assessed by two different physiotherapist observers. The timed 360° turn test, Expanded and revised Gross Motor Function Classification System (GMFCS-E&R) for functional motor levels of the subjects, lower extremity muscle tone will be measured with the Modified Ashworth Scale (MASH) at the beginning of the one-time study and recorded. Pediatric Berg Balance Scale, Timed Up and Go Test, Pediatric Functional Reaching test and Modified Four Square Stepping Test, 3m walking back test (3MGYT) will be performed.Evaluations will be made by two separate physiotherapists with at least 5 years of experience in this field. The time it took for individuals to complete activities during the tests with a stopwatch will be recorded.
  Other Names: the timed 360° turn test

SUMMARY:
Cerebral Palsy (CP) is a non-progressive neurodevelopmental disorder that starts in the early stages of life, causes activity limitation, and consists of movement and posture deficiencies. Children with CP usually have difficulties in mobility, transfer and social participation due to many motor and sensory disorders such as muscle weakness, decreased postural control, balance, spasticity. Many children with CP have difficulty in balancing independently, walking, walking on hills/uneven ground, and performing daily physical functions.

DETAILED DESCRIPTION:
Abnormal gait patterns and balance problems are common problems in children with CP. As children get older, these impairments in walking abilities become more pronounced. In addition to all these problems, hypertonus, increased stretch reflex, muscle weakness, coactivation of antagonist muscles, posture disorders, proprioception losses, muscle and joint deformities are other factors that cause gait disorders and balance problems in children with CP. At this point, the main purpose of CP rehabilitation is to ensure that the child gains maximum functional independence by achieving optimal developmental potential. Therefore, balance and gait restrictions are important problems in children with CP. For these reasons, the evaluation of gait and balance is of great importance in terms of determining the effectiveness of the physiotherapy program, shaping the program, planning and determining the effectiveness of orthopedic and surgical applications, especially in children with CP who have walking potential. In the literature, gait pathologies in children with CP and easy-to-use, valid and reliable observational gait analyzes that can evaluate gait in the clinic are emphasized.Gait analysis systems including computerized kinetics and kinematics laboratories, electromyography (EMG) and video imaging are the "gold standard" methods used to evaluate the gait of children with CP. However, these evaluation methods are not routinely used in clinics because they are complex, expensive, time-consuming and not easy to apply. In addition to many gait assessment scales, the standing, walking, running and stair climbing sections of Gross Motor Function Measurement (GMFM) are widely used in the clinic to evaluate gait. In addition to all these, performance tests that are commonly used in the clinic, such as the Timed Sit and Go Test, the Up and Down Stair Climbing Test, the 2 Minute Walk Test, and the 6 Minute Walk Test, evaluate the functionality of gait. All these tests are tests that evaluate gait prospectively and cannot fully address the functional status of the child. Therefore, in order to gain and maintain functional independence, the gait problems of the child with CP need to be examined more. In this respect, it provides a different task than normal with the evaluation of rotation, allowing the observation of body perception, trunk stability, balance, correction and protective reactions provided by anterior-posterior cocontraction. This observation can provide the exact determination of the problem that will guide the treatment. The timed 360° turn test is a standard clinical measure used to evaluate dynamic standing balance. When the literature was reviewed, no study was found about the The timed 360° turn test in children with CP. The aim of the study is to examine the validity and reliability of The timed 360° turn test in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with CP according to SCPE criteria
* Level ≤ 2 by GMFCS-E&R
* Children aged 7-18 with CP with a Communication Function Classification System (CFCS) ≤ 3
* Children with a Modified Ashworth Scale (MASH) ≤ 3
* Passive range of motion in the ankle, knee and hip joints
* Individuals with spastic hemiparetic-diparetic CP who can follow verbal commands
* Volunteer to participate in the study

Exclusion Criteria:

* Have not had Botox, (Botulinum toxin) or surgery in the last 6 months
* Contracture of ankle and knee joint
* Individuals with hemiparetic-diparetic CP who can follow verbal commands

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with spastic diparetic and hemiparetic cerebral palsy
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
the timed 360° turn test | two different observers' measurements in 2 different days (2 sessions per day on two separate days)
  In the timed 360° turn test, any marker, such as a tape or pen, is used to determine the starting point and a stopwatch is used to measure time. Each participant stands up comfortably at the starting point and rotates 360° for both sides. The time begins with the word "begin" and ends when the participants' shoulders look forward again. Each participant completes. The average of 3 trials and 3 trials for each side yields a result. The average score is recorded for the timed 360° turn test performance.
Four Square Step Test (FSST) | first day of assessment
  The child stands in square 2 facing square 1 in a marked area divided into 4 squares. The child has to take turns stepping on each square as fast as possible: it requires the child to step forward, backward, right, and left in a sequence of 2, 3, 4, 1, 4, 3, 2, and 1, respectively. The necessary equipment is a stopwatch and 4 walking sticks 90 cm long. A square with 4 is formed by laying the canes flat on the ground. If the child cannot complete the series, loses balance or touches the cane during the trial, the trial is repeated.Two FSSTs are completed with the best time taken as a score.Timing begins with the first foot touching the floor in frame 1 and ends with the last foot touching the floor in frame 4. Test performance is measured in seconds (sec) and shorter completion time means better dynamic stability.
Pediatric Berg Balance Scale (PBBS) | first day of assesment
  The test has 14 items of increasing difficulty to test functional skills related to activities of daily living, from sitting to standing on one leg. Each item is scored on a five-point ranking scale ranging from 0 to 4 points, with a maximum score level of 56. A higher score indicates better postural balance.
Timed Up and Go Test (TUG) | first day of assesment
  For the test, the child is seated in a height-adjustable chair. The chair height is adjusted so that the child's feet are in contact with the floor and the knees and hips are flexed to 90 degrees. A distance of 3 meters is marked. When the command is given, the child is asked to get up, walk, return and sit on the chair until the marked area. By starting the time with the start command, the time until sitting is recorded. This test will be repeated 3 times and the average time will be recorded. Increasing time indicates worse dynamic stability.
Pediatric Functional Reach test | first day of assesment
  The child is asked to stand sideways on a wall, with the elbows extended at 90 degrees of shoulder flexion without touching the wall. The first measurement is made in this position. Then, he is asked to reach forward without taking a step. The last point it can reach is recorded. The distance between these two distances is measured in meters and recorded. The test is repeated when stepping or stopping the contact of the foot with the ground. A higher measurement indicates worse balance.

SECONDARY OUTCOMES:
Expanded and revised Gross Motor Function Classification System (GMFCS-E&R) | first day of assessment
  It is a standard classification system used to classify gross motor functions of children with CP. GMFCS-E&R classifies levels I to V. Level I indicates the best and V the worst level of motor function.
Modified Ashworth Scale (MASH) | first day of assessment
  It is a method used to determine the severity of spasticity. It is based on the subjective rating of the resistance felt during the examination. Spasticity of the bilateral hip adductors, hip flexors, knee flexors, ankle plantar flexors (gastro-solues) muscles in the lower extremity will be evaluated once at the beginning of the treatment program. The tone felt in these muscles against passive movement is classified as follows; 0: No increase in tone, 1: Slight increase in tone characterized by catching and relaxation or mild resistance at the end of the ROM, 1+: Slight increase in tone characterized by minimal resistance in the remaining ROM (less than half) after capture, 2: Significant tone over most of the ROM increase, but the involved joint can be moved easily, 3: Significant increase in muscle tone, passive movement is difficult, 4: The involved part is rigid in flexion or extension.
Demographic information of the children | first day of assessment
  age, height, gender, education level, background of physiotherapy and diagnosis will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No